CLINICAL TRIAL: NCT05170711
Title: the Effect of Hypotensive Anesthesia With Sleeve Gastrectomy
Brief Title: Hypotensive Anesthesia With Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant professor & consultant of general surgery, Department of Surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fac.med 21.50
Record Dates: First submitted 2021-12-11; First posted 2021-12-28 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypotensive anesthesia (Experimental): hypotensive anesthesia group
  Interventions: Procedure: hypotensive anesthesia
- normotensive anesthesia (Active Comparator): normotensive anesthesia group
  Interventions: Procedure: normotensive anesthesia

INTERVENTIONS:
Procedure: hypotensive anesthesia — hypotensive anesthesia
  Arms: hypotensive anesthesia
Procedure: normotensive anesthesia — normotensive anesthesia group
  Arms: normotensive anesthesia

SUMMARY:
to do sleeve gastrectomy under hypotensive anesthesia till compete stapling then hypertensive at the end

DETAILED DESCRIPTION:
to do sleeve gastrectomy under hypotensive anesthesia till compete stapling then hypertensive at the end of the operation to check bleeding

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 or more than 35 with comorbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 50
* patients with BMI less than 35
* patient with previous upper abdominal surgery either for obesity or other diseases
* patients with GERD

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
operative time | 20-120 minutes
  operative time from skin to skin
intraoperative bleeding or oozing | 0-120 minute
  intraoperative bleeding or oozing by the number of used gauzes and clips

SECONDARY OUTCOMES:
postoperative bleeding | 2-36 hours
  the incidence of postoperative bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Minya, Egypt